CLINICAL TRIAL: NCT05799261
Title: Clinical Evaluation of a Novel Protocol (Guided Biofilm Management) for Supportive Periodontal Therapy: a Long-term Randomized Controlled Clinical Study
Brief Title: Novel Protocol for Supportive Periodontal Therapy
Acronym: GBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-00046
Record Dates: First submitted 2022-12-23; First posted 2023-04-05 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis
Keywords: Guided biofilm management; Supportive periodontal therapy
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Patients in supportive periodontal therapy will be treated according to standard protocols of the Department of Periodontology. The test group patient will undergo treatment by the concept of Guided Biofilm Management consisting of removal of soft supra- and subgingival bacterial deposits by means of erythritol powder air-polishing, followed by the local precise removal of hard deposits and a subsequent use of another sub- and supragingival erythritol powder air-polishing. The study duration will be 3 years.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (standard protocol) (Active Comparator): The control group will be treated according to standard protocols of the Department of Periodontology of the university of Bern and receive conventional scaling and root planing. Supra- and subgingival hard and soft tissue deposits are being removed by means of hand instruments and ultra-sonic scalers followed by rubber cup polishing. All patients will have 2 visits per year. At each visit outcome measures will be assessed by masked dentists.
  Interventions: Procedure: Control (standard protocol)
- Test (Guided Biofilm management) (Experimental): The test group will be treated according to a novel treatment concept (Guided biofilm management, GBM):
  1. Staining of all tooth surfaces to detect soft and hard deposits.
  2. Removal of supra- and subgingival hard and soft bacterial deposits by means of an erythritol powder air-polishing.
  3. If present, the supra- and subgingival hard deposits (e.g. calculus) will be removed by means of a slim ultrasonic tip (Piezon PS, EMS, Nyon Switzerland) without any additional use of hand instruments.
  4. Another sub- and supragingival application of erythritol powder air-polishing without any rubber cup polishing. All patients will have 2 visits per year. At each visit outcome measures will be assessed by masked dentists.
  Interventions: Procedure: Test (Guided Biofilm management)

INTERVENTIONS:
Procedure: Control (standard protocol) — The control group will be treated according to standard protocols of the Department of Periodontology of the university of Bern and receive conventional scaling and root planing. Supra- and subgingival hard and soft tissue deposits are being removed by means of hand instruments and ultra-sonic scalers followed by rubber cup polishing. All patients will have 2 visits per year. At each visit outcome measures will be assessed by masked dentists.
  Arms: Control (standard protocol)
Procedure: Test (Guided Biofilm management) — The test group will be treated according to a novel treatment concept (Guided biofilm management, GBM):
  1. Staining of all tooth surfaces to detect soft and hard deposits.
  2. Removal of supra- and subgingival hard and soft bacterial deposits by means of an erythritol powder air-polishing.
  3. If present, the supra- and subgingival hard deposits (e.g. calculus) will be removed by means of a slim ultrasonic tip (Piezon PS, EMS, Nyon Switzerland) without any additional use of hand instruments.
  4. Another sub- and supragingival application of erythritol powder air-polishing without any rubber cup polishing. All patients will have 2 visits per year. At each visit outcome measures will be assessed by masked dentists.
  Arms: Test (Guided Biofilm management)

SUMMARY:
Supportive periodontal therapy (SPT) succeeds the active phase of periodontal therapy. SPT includes repeated supra- and subgingival scaling and root planing (SRP) at all sites with bleeding on probing and pocket depths ≥ 4-5 mm. Despite the fact that this treatment approach has been proven to be extremely successful, on a long-time basis, it is associated with substantial hard tissue loss (i.e. root cementum and dentin) that may lead to an increase in hypersensitivity, weakening of the tooth and even endodontic complications. Therefore, a novel treatment concept (Guided Biofilm Management or GBM) consisting of removal of all soft supra- and subgingival bacterial deposits by means of an erythritol powder air-polishing, followed by the local, precise removal of supra and subgingival hard deposits (e.g. calculus) and subsequent use of another sub- and supragingival erythritol powder air-polishing, has been introduced. Here, the investigators will compare this novel concept (GBM) with the conventional care during SPT using hand curettes.

DETAILED DESCRIPTION:
There is solid scientific evidence demonstrating that the clinical results obtained following active periodontal therapy can be maintained on a long-term basis provided that regular supportive periodontal therapy (SPT) is rendered. On a routine basis, SPT includes repeated supra- and subgingival scaling and root planing (SRP) at all sites with bleeding on probing and pocket depths ≥ 4-5 mm. Despite the fact that this treatment approach has been proven to be extremely successful, on a long-time basis, it is associated with substantial hard tissue loss (i.e. root cementum and dentin) that may lead to an increase in hypersensitivity, weakening of the tooth and even endodontic complications. Since patients enrolled in SPT have usually probing pocket depths (PPD) < 6 mm and limited supra- and subgingival deposits, the question arises whether SRP by means of hand and ultrasonic instruments may be needed at all sites with a PPD > 4 mm with BOP (+) that do not exhibit hard bacterial deposits (e.g. supra and subgingival calculus). It has been repeatedly shown that bacterial deposits can be removed from the root surfaces by mere polishing without any SRP, thus leading to comparable clinical outcomes than following the use of conventional SRP by means of hand instruments (e.g. metal curettes). The removal of "diseased" root cementum is therefore not necessary to accomplish clinical success. Results from a recent "in-vitro" study using a novel "subgingival pocket model" have shown that compared to hand instrumentation, the application of an air-polishing with erythritol prevents substance-loss and results in a smooth surface with nearly no residual biofilm that promotes the reattachment of PDL fibroblasts. These findings are in line with the results of a randomized controlled clinical study which has shown that biofilm removal by means of an erythritol powder based air-polishing yielded similar outcomes to those obtained with conventional SRP. Moreover, the use of the erythritol powder air-polishing yielded statistically and clinically better patient acceptance.

Based on these results a novel treatment concept (Guided Biofilm Management or GBM) consisting of removal of all soft supra- and subgingival bacterial deposits by means of an erythritol powder air-polishing, followed by the local, precise removal of supra- and subgingival hard deposits (e.g. calculus) and subsequent use of another sub and supragingival erythritol powder air-polishing, has been introduced.

The authors hypothesize that this approach may enable to render a more personalized and precise treatment for patients enrolled in SPT, thus leading to less hard tissue loss and better patient acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient adherent to supportive periodontal therapy
* With < 6 mm probing pocket depth (PPD)

Exclusion Criteria:

* Clinically significant concomitant diseases
* Enrolment in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Change in bleeding on probing | Over the study period of 3 years at every recall (i.e. every 6 months)
  This is a categorical variable defined as the percentage of bleeding sites out of the total number of sites. Hereby, all gingival sulci and pockets will be measured with a periodontal probe and bleeding sites will be recorded. The maximum is 100% and the minimum 0%. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Change in probing pocket depth | Over the study duration of 3 years at every recall (i.e. every 6 months)
  Pocket depths will be measured by means of a periodontal probe. The minimal clinically measured pockets are 1 mm and the maximal value for pocket depths allowed in this study is 5 mm. Higher pocket depth values represent worse results. With respect to the reduction in probing depth it is the other way round. A higher value of 3 mm (maximal reduction value) represent better outcomes and a smaller reduction or none (0 mm).
Clinical attachment level | At the beginning of the study, after 1 year and after 3 years
  Gingival recessions and pockets depths both measured with millimeter-indicating periodontal probes will be measured and added to the clinical attachment loss/level. Minimal values are 0 mm or even 1 to 2 mm below zero. While maximal values are around 3 mm.
Patient comfort | Over the study duration after 1, 2, and 3 years
  Assessed by a Visual Analogue Scale (VAS). VAS is a 100 mm scale with 0 being the worst imaginable satisfaction and 100 mm perfect satisfaction with the treatment. In terms of pain it is the opposite with 0 representing no pain and 100 mm the worst imaginable pain sensation.
Time effectiveness | Over the study duration of 3 years at every recall (i.e. every 6-months)
  The time that is needed to do a thorough cleaning according to the respective protocol the patient was allocated to. For this purpose the dental hygienists are recording the time in minutes. Minimal amount of time is 30 minutes and maximal time is 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Sculean, Prof., Principal Investigator — University of Bern
Locations (1):
- Department of Periodontology, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Hagi TT, Hofmanner P, Eick S, Donnet M, Salvi GE, Sculean A, Ramseier CA. The effects of erythritol air-polishing powder on microbiologic and clinical outcomes during supportive periodontal therapy: Six-month results of a randomized controlled clinical trial. Quintessence Int. 2015 Jan;46(1):31-41. doi: 10.3290/j.qi.a32817. PMID 25262675
- [Result] Hagi TT, Klemensberger S, Bereiter R, Nietzsche S, Cosgarea R, Flury S, Lussi A, Sculean A, Eick S. A Biofilm Pocket Model to Evaluate Different Non-Surgical Periodontal Treatment Modalities in Terms of Biofilm Removal and Reformation, Surface Alterations and Attachment of Periodontal Ligament Fibroblasts. PLoS One. 2015 Jun 29;10(6):e0131056. doi: 10.1371/journal.pone.0131056. eCollection 2015. PMID 26121365
- See also: Standardized human dentin specimens were colonized by multi-species biofilms for 3.5 days and subsequently treated as follows: a) hand-instrumentation b) ultrasonication c) air-polishing using erythritol and d) erythritol combined with chlor — https://pubmed.ncbi.nlm.nih.gov/26121365/
- See also: 40 chronic periodontitis patients previously enrolled in SPT were randomly assigned into two groups for the treatment with subgingival EPAP or repeated scaling and root planing (SRP). — https://pubmed.ncbi.nlm.nih.gov/25262675/